CLINICAL TRIAL: NCT00696332
Title: A Multinational, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Tolerability and Safety of Talampanel in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Talampanel for Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALS-TAL-201 (ALSTAR); ALSTAR
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: ALS
Keywords: ALS
MeSH Terms: interventions — talampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Talampanel 50mg (Experimental): 50mg Talampanel 3 times per day
  Interventions: Drug: Talampanel
- Talampanel 25mg (Experimental): 25mg Talampanel 3 times per day
  Interventions: Drug: Talampanel
- Placebo (Placebo Comparator): placebo 3 times per day
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Talampanel — capsules Talampanel, 3 times per day, 52 weeks
  Other Names: AMPA antagonist
  Arms: Talampanel 50mg
Drug: Talampanel — capsules Talampanel, 3 times per day, 52 weeks
  Other Names: AMPA antagonist
  Arms: Talampanel 25mg
Other: placebo — capsules, placebo, 3 times a day, for 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, tolerability and safety of oral administration of talampanel compared to a placebo in subjects with ALS.

ELIGIBILITY:
Subjects with sporadic or familial ALS classified as definite, probable, or laboratory-supported probable ALS according to the revised El Escorial criteria.

Inclusion Criteria:

1. Diagnosis of definite or probable ALS in accordance with the El-Escorial criteria.
2. Subject has experienced his/her first ALS symptoms within 3 years prior to the screening visit.
3. Slow VC test equal to or greater than 70% of the predicted value.
4. The sum of the 3 respiratory items on the ALSFRS-R must total at least 10 points.
5. Subjects taking riluzole must be on a stable dose for at least 8 weeks prior to screening visit.
6. Ages 18-80 (inclusive)

Exclusion Criteria:

1. The use of invasive or non-invasive ventilation.
2. Subject having undergone gastrostomy.
3. Subject with any clinically significant or unstable medical condition.
4. Subject participating in any other investigational drug trial or using investigational drug (within 12 weeks prior to screening and thereafter).
5. Females who are pregnant or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in ALS Functional Rating Score (ALSFRS-R slope) | 52 weeks

SECONDARY OUTCOMES:
Time from baseline to the first occurrence of either death, tracheostomy or permanent assisted ventilation. | 52 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- United States (7):
  - CA Medical Center for Movement Disorders-Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Kansas Medical Center - Dept of Neurology, Kansas City, Kansas
  - Johns Hopkins OPC - Meyer Bldg, Baltimore, Maryland
  - Massachusetts General Hospital-Neurology Clinical Trials Unit, Charlestown, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University - Neurology Institute, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
- Academic Hospital University of Leuven - ALS dept, Leuven, Belgium
- Canada (3):
  - ALS Centre, Vancouver, British Columbia
  - London Health Sciences Centre Motor Neuro Diseases Clinic, London, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- France (3):
  - C.H.U. La Timone - Service de Neurologie, Marseille
  - C.H.U. de Montpellier - Hopital Gui de Chauliac - Service des Explorations Neurologiques, Montpellier
  - Hopital La Pitie Salpetriere - Federation de Neurologie, Paris
- Germany (3):
  - Universitaetsklinik Berlin-Charite, Campus Virchow Klinikum, Neurologische Klinik, Berlin
  - Berufsgenossenschaftliche Klinik Bergmannsheil, Neurologische Klinik, Bochum
  - Universitaet Ulm, Ulm
- Semmelweis University, Department of Neurology, Budapest, Hungary
- Sourasky MC -EMG Unit, Tel Aviv, Israel
- Italy (3):
  - Fondazione "S.Maugeri" Clinica della Riabilitazione IRCCS-Istituto Scientifico di Lissone, Lissone (MI)
  - Centro Clinico NEMO, Milan
  - Azienda Ospedaliero Universitaria San Giovanni Battista di Torino - Dipartimento di Neuroscienze, Torino
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Carlos III, Madrid, Spain